CLINICAL TRIAL: NCT04691674
Title: Optimal Placement Duration of Pancreatic Duct Stent Inserted During ERCP: 2 vs 4 Weeks
Brief Title: Optimal Placement Duration of Pancreatic Duct Stent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DongGuk University (Other)
Collaborators: Seoul National University Hospital (Other); Gachon University Gil Medical Center (Other); Gyeongsang National University Hospital (Other); Kyungpook National University Hospital (Other); Severance Hospital (Other); The Catholic University of Korea (Other); Korea University Ansan Hospital (Other); Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Kee Jang, Principal investigator, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-10-024-003
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cholangitis; Post-ERCP Acute Pancreatitis; Stent Dislodgement
MeSH Terms: conditions — Cholangitis | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Endoscopic removal of pancreatic duct stent at 4 weeks following ERCP, unless spontaneously dislodged.
  Interventions: Procedure: Endoscopy
- Control group (Placebo Comparator): Endoscopic removal of pancreatic duct stent at 2 weeks following ERCP, unless spontaneously dislodged.
  Interventions: Procedure: Endoscopy

INTERVENTIONS:
Procedure: Endoscopy — Endoscopic removal of the pancreatic stent

SUMMARY:
A randomized controlled trial to determine the optimal placement duration of pancreatic duct stents (PDS) inserted during ERCP: 2 vs 4 weeks

DETAILED DESCRIPTION:
Endoscopic pancreatic duct stenting has been increasingly used for the treatment of a variety of pancreatic disorders including chronic pancreatitis, pancreatic duct stricture, drainage of pseudocysts, and the prevention of pancreatitis following endoscopic retrograde cholangiopancreatography (ERCP). Several randomized, controlled trials and meta-analyses have proven a significant reduction in incidence and severity of post-ERCP pancreatitis (PEP) with prophylactic pancreatic duct stenting. The US and European guidelines recommend that pancreatic duct stents (PDS) be placed between 7-10 days and 5-10 days, respectively, in order to prevent PEP in some situations. Therefore, the placement of PDS has been an established essential procedure for preventing a fatal complication, PEP. Furthermore, PDS placement can facilitate difficult common bile duct cannulation. It may help not only to straighten papillary anatomy but also to identify the location of the biliary orifice.

However, PDS tends to become occluded easily due to protein content, calcium carbonate crystals, and bacteria in the pancreatic juice. The occluded PDS can cause acute pancreatitis or abdominal pain. For this reason, the guidelines recommend PDS be placed within 10 days. Because of this policy, the patient must take the inconvenience of undergoing another endoscopic procedure to remove the PDS. However, all patients with occluded PDS do not have symptoms such as pain. In one series, only 6 percent of patients with clogged PDS developed symptoms. The low incidence of symptoms despite a high rate of stent occlusion suggests that the stent may function as a wick around which pancreatic juices continue to drain. In addition, the rate of spontaneous stent dislodgement was relatively high (65-86%) within 30 days according to a previous study. A recent study also reported that prolonged retention of prophylactic pancreatic stents is not associated with increased complications.

Taken together, PDS placed during ERCP do not need to be removed until any symptom develops. In particular, if the investigators can observe PDS for about a month without removing them, the PDS are more likely to pass out spontaneously, which could reduce unnecessary procedures. However, to date, there have been few randomized controlled studies on the optimal placement duration of PDS inserted during ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent the pancreatic duct stent placement during ERCP

Exclusion Criteria:

* Patients who had pancreatic duct stent for the purpose of pancreatic interventions
* Patients who underwent simultaneous bile duct stenting

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with undergoing endoscopic procedures | 2 weeks (control group) or 4 weeks (study group) following ERCP
  The necessity of endoscopic procedure for pancreatic duct stent removal

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mazaki T, Mado K, Masuda H, Shiono M. Prophylactic pancreatic stent placement and post-ERCP pancreatitis: an updated meta-analysis. J Gastroenterol. 2014 Feb;49(2):343-55. doi: 10.1007/s00535-013-0806-1. Epub 2013 Apr 24. PMID 23612857
- [Result] Choudhary A, Bechtold ML, Arif M, Szary NM, Puli SR, Othman MO, Pais WP, Antillon MR, Roy PK. Pancreatic stents for prophylaxis against post-ERCP pancreatitis: a meta-analysis and systematic review. Gastrointest Endosc. 2011 Feb;73(2):275-82. doi: 10.1016/j.gie.2010.10.039. PMID 21295641
- [Result] ASGE Standards of Practice Committee; Chandrasekhara V, Khashab MA, Muthusamy VR, Acosta RD, Agrawal D, Bruining DH, Eloubeidi MA, Fanelli RD, Faulx AL, Gurudu SR, Kothari S, Lightdale JR, Qumseya BJ, Shaukat A, Wang A, Wani SB, Yang J, DeWitt JM. Adverse events associated with ERCP. Gastrointest Endosc. 2017 Jan;85(1):32-47. doi: 10.1016/j.gie.2016.06.051. Epub 2016 Aug 18. No abstract available. PMID 27546389
- [Result] Dumonceau JM, Kapral C, Aabakken L, Papanikolaou IS, Tringali A, Vanbiervliet G, Beyna T, Dinis-Ribeiro M, Hritz I, Mariani A, Paspatis G, Radaelli F, Lakhtakia S, Veitch AM, van Hooft JE. ERCP-related adverse events: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2020 Feb;52(2):127-149. doi: 10.1055/a-1075-4080. Epub 2019 Dec 20. PMID 31863440
- [Result] Goldberg E, Titus M, Haluszka O, Darwin P. Pancreatic-duct stent placement facilitates difficult common bile duct cannulation. Gastrointest Endosc. 2005 Oct;62(4):592-6. doi: 10.1016/j.gie.2005.04.046. PMID 16185975
- [Result] Deviere J. Why do pancreatic stents become occluded? Gastrointest Endosc. 2005 Jun;61(7):867-8. doi: 10.1016/s0016-5107(05)00548-1. No abstract available. PMID 15933689
- [Result] Ikenberry SO, Sherman S, Hawes RH, Smith M, Lehman GA. The occlusion rate of pancreatic stents. Gastrointest Endosc. 1994 Sep-Oct;40(5):611-3. doi: 10.1016/s0016-5107(94)70264-0. No abstract available. PMID 7988829
- [Result] Rashdan A, Fogel EL, McHenry L Jr, Sherman S, Temkit M, Lehman GA. Improved stent characteristics for prophylaxis of post-ERCP pancreatitis. Clin Gastroenterol Hepatol. 2004 Apr;2(4):322-9. doi: 10.1016/s1542-3565(04)00062-x. PMID 15067627
- [Result] Dultz G, Gerber L, Zeuzem S, Bojunga J, Friedrich-Rust M. Prolonged retention of prophylactic pancreatic stents is not associated with increased complications. Pancreatology. 2019 Jan;19(1):39-43. doi: 10.1016/j.pan.2018.11.011. Epub 2018 Nov 22. PMID 30502123